CLINICAL TRIAL: NCT05980390
Title: Assessment of Tissue Levels of IL-35 in Active and Stable Vitiligo
Brief Title: IL35 Level in Vitiligo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dr, Cairo University
Other Study IDs: IL35 in vitiligo
Record Dates: First submitted 2023-07-29; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: IL35, Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active vitiligo
  Interventions: Diagnostic Test: IL 35 in tissue biopsy
- Stable vitiligo
  Interventions: Diagnostic Test: IL 35 in tissue biopsy
- Normal controls
  Interventions: Diagnostic Test: IL 35 in tissue biopsy

INTERVENTIONS:
Diagnostic Test: IL 35 in tissue biopsy — Elisa testing

SUMMARY:
The aim of this observational study is to evaluate the level of the IL-35 protein in tissue biopsy from patients with active & stable vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active and stable vitiligo

Exclusion Criteria:

* Pregnant and lactating women.
* Patients with associated autoimmune or other dermatological diseases e.g., Alopecia areata and lupus erythematous.
* Patients already on both topical and systemic treatment at the time of recruitment.
* Patients on Immunosuppressive drugs.
* Other hypopigmented diseases such as pityriasis alba, tinea versicolor, lichen sclerosis, post inflammatory hypopigmentation and leprosy as excluded by lack of accentuation by wood's light examination.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients with active and stable vitiligo together with normal subjects
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
level of IL35 in tissue biopsy | 3 months